CLINICAL TRIAL: NCT02853799
Title: Comparison of the Effects of Intermittent and Continuous Enteral Feeding on Glucose-Insulin Dynamics in Critically Ill Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tyson Sjulin, D.O., Pulmonary/Critical Care Fellow, San Antonio Military Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: x5tjqsc6
Record Dates: First submitted 2016-07-21; First posted 2016-08-03 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Glucose-insulin Dynamics
MeSH Terms: interventions — Osmolite; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Enteral Feeding (Other): Crossover Study:
  Randomized to continuous enteral feeding first then crossed over to receive versus intermittent enteral feeding next.
  Interventions: Other: Comparison of the Effects of Intermittent and Continuous Enteral Feeding on Glucose-Insulin Dynamics in Critically Ill Medical Patients; Dietary Supplement: Osmolite 1.2 cal/ml Enteral Feeds
- intermittent enteral feeding (Other): Crossover Study:
  Randomized to intermittent enteral feeding first then crossed over to receive versus continuous enteral feeding next.
  Interventions: Other: Comparison of the Effects of Intermittent and Continuous Enteral Feeding on Glucose-Insulin Dynamics in Critically Ill Medical Patients; Dietary Supplement: Osmolite 1.2 cal/ml Enteral Feeds

INTERVENTIONS:
Other: Comparison of the Effects of Intermittent and Continuous Enteral Feeding on Glucose-Insulin Dynamics in Critically Ill Medical Patients — 1. Placement of feeding tube stomach (oral- or naso-gastric tube)
  2. Randomized to receive either continuous feeding or intermittent feeding first. Once at goal nutrition for 4 hours, enter first 4-hour data collection interval. Next proceed with cross-over and complete a 4-hour washout period with the feed type. Finally enter second 4-hour data collection period. To enter into the first data collection period, the patient would require an insulin infusion.
  3. There will be five blood glucose checks in each data collection period.
  4. If two blood glucose concentrations are above 180 mg/dl then a regular insulin infusion will be initiated.
Dietary Supplement: Osmolite 1.2 cal/ml Enteral Feeds — Osmolite 1.2 cal/ml Enteral Feeds via feeding tube (oral- or naso-gastric tube)

SUMMARY:
Continuous enteral feeding is the most common type of nutrition used in critically ill patients despite being non-physiologic, as all mammalian alimentary tracts have been designed for intermittent ingestion of nutrients. The small numbers of randomized controlled studies that have compared intermittent gastric feeds (IGF) to continuous gastric feeds (CGF) in intensive care units have demonstrated that IGF is safe, feasible and have the shorter time to goal nutrition. Studies of healthy adults have also demonstrated that the mean glucose concentration (MGC) is lowered when bolus enteral feedings are used instead of continuous feeds; these changes in glucose-insulin metrics might be beneficial to a critically ill patient population where stress hyperglycemia is common. This study will compare the effects of CGF and IGF in a critically ill medical patient population. Glucose-insulin dynamics for each type of enteral feed will be analyzed by performing a randomized crossover study to compare the effects of CGF and IGF on MGC, total insulin infused, glucose variability (GV), episodes of hypoglycemia and maximum glucose concentration values.

DETAILED DESCRIPTION:
This will be a non-blinded randomized crossover study in a generalized population of critically ill adults. The population of this study is defined from the ages of 18-90 admitted to the Medical Intensive Care Unit (MICU). This study will compare the glucose-insulin dynamics in critically ill adults that are feed using either a CGF or IGF scheme while their glucose concentrations are maintained between 140-180 mg/dl using an insulin infusion protocol. Randomization performed using computer generated random numbers kept individually in sealed envelopes. All participants will have nasal gastric or oral gastric (NG/OG) tube previously placed for their nutritional needs. The amount of Osmolite given will be determined by the ideal weight for each participant: 1.2 cal/ml Osmolite with caloric goal of 25 kcal/kg/day. Feeding intolerance develops which is defined as: excessive abdominal distention, emesis, abdominal pain, vomiting and gastric residual > 250 ml for IGF and gastric residual > 500 ml for CGF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Anticipated ICU stay greater than 72 hours
* Expected indication for enteral feeding within first 24-48 hours of ICU admission

Exclusion Criteria:

* Any contraindications relating to an oral or nasal gastric tube, Osmolite 1.2 cal/ml, goal rate (or goal volume) of Osmolite 1.2 cal/ml using a 24-hour goal nutrition, gastric feeds due to anatomical/physiological pathology, ideal body weight that exceeds 85 kg to maintain goal volumes in the intermittent arm below 301 ml or a potassium greater than 6.4.
* Planned procedures or tests that would require holding gastric feeds during the protocol.
* Pregnancy, confirmed by pregnancy test on all females < 60 years of age.
* Hemodynamic instability as defined by any vasoactive medication requirement for blood pressure support or cardiac arrhythmias to include: Norepinephrine ≥ 5 mcg/min, Epinephrine ≥ 5 mcg/min, Dopamine > 5 mcg/kg/min, Milrinone 0.375mcg/kg/min, Vasopressin > 0.04 Units/min, Dobutamine > 5 mcg/kg/min, any other vasoactive drip, and any combination of low dose vasopressors listed above. Atrial Nodal blocking agents used in a continuous drip form to include diltiazem, esmolol and amiodarone are allowed if not requiring the above vasoactive medications restrictions.
* Prior surgical procedure that would preclude a goal rate/or volume for CGF/IGF to include: previous partial or complete gastrectomy or massive intestinal resection leaving less than 200 cm of small bowel.
* Screening glucose concentration less than 120 mg/dl while NPO unless diabetic.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Total insulin infused | total time in the protocol should be 36 hours to include crossover
  Total insulin infused

SECONDARY OUTCOMES:
Mean glucose concentration | time the protocol should be 36 hours to include crossover
  Mean glucose concentration

OTHER OUTCOMES:
Glucose standard deviation | total time in the protocol should be 36 hours to include crossover
  Glucose standard deviation
Maximum glucose concentration | total time in the protocol should be 36 hours to include crossover
  Maximum glucose concentration
Minimum glucose concentration | total time in the protocol should be 36 hours to include crossover
  Minimum glucose concentration
Episodes of hypoglycemia | total time in the protocol should be 36 hours to include crossover
  Glucose concentration < 70 mg/dl

REFERENCES:
- Available data/document: Study Protocol — http://journals.lww.com/annalsofsurgery/pages/articleviewer.aspx?year=2016&issue=03000&article=00007&type=abstract — 2. Chowdhury, Abeed H., et al. "Effects of Bolus and Continuous Nasogastric Feeding on Gastric Emptying, Small Bowel Water Content, Superior Mesenteric Artery Blood Flow, and Plasma Hormone Concentrations in Healthy Adults: A Randomized Crossover Study." Annals of Surgery (2014).